CLINICAL TRIAL: NCT05379933
Title: C-PRIME: Caregiver Protocol for Remotely Improving, Monitoring, and Extending Quality of Life
Brief Title: Caregiver Protocol for Remotely Improving, Monitoring, and Extending Quality of Life
Acronym: C-PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-21751
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Stress; Quality of Life; Sleep Disturbance
Keywords: Family Caregiver; Well-being
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-PRIME (Experimental): Participants will wear an activity tracker for 8 weeks. During the 8 weeks of the study, participants will complete weekly survey questions about health and well-being and engage in weekly, 15-20 minute telephone/videoconference coaching sessions with a health coach.
  Interventions: Other: Remote health coaching to improve self-care behaviors

INTERVENTIONS:
Other: Remote health coaching to improve self-care behaviors — Participants will be asked to wear an activity tracker, complete brief surveys, and participate in weekly health coaching sessions remotely for 8 weeks

SUMMARY:
The purpose of this study is to test an intervention to improve health promoting behaviors in family caregivers of patients receiving cancer therapy

ELIGIBILITY:
Inclusion Criteria:

* Eligible family caregivers will be:
* An unpaid family member or friend who provides assistance and support with healthcare of a non-institutionalized patient receiving some form of treatment for stage III or IV colorectal cancer at Moffitt Cancer Center
* Age 18+ years
* English or Spanish speaking
* Able to complete questionnaires and engage in short discussions with coaches
* Able to identify a primary care medical provider
* Willing/able to use a mobile device provided by the study team or their own their device.

Exclusion Criteria:

* Participants who do not meet the study inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Agree to Participate (Acceptability) | 12 Months
  The study will be deemed acceptable if at least 50% of eligible family caregivers agree to participate
Percentage of Participants Who Provide Data (Feasibility) | 12 Months
  The study will be deemed feasible if at least 75% of family caregivers who participate provide data for at least 50% of study days

SECONDARY OUTCOMES:
Self Care Behaviors - Primary Efficacy | 8 Weeks
  Participant's self care behaviors will be measured using the Health-Promoting Lifestyle Profile-II. This is a 52-item questionnaire that assesses use of behaviors likely to promote a healthy lifestyle and indicate greater selfcare. Responses are categorized into an overall health-promoting lifestyle score as well as subscales assessing health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations, and stress management.
Quality of Life -Secondary Efficacy | 8 Weeks
  Participants' quality of life will be assessed using the EORT QLQ-C30, a 30-item measure that assesses quality of life in various domains of functioning and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Gonzalez, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gudenkauf LM, Li X, Hoogland AI, Oswald LB, Lmanirad I, Permuth JB, Small BJ, Jim HSL, Rodriguez Y, Bryant CA, Zambrano KN, Walters KO, Reblin M, Gonzalez BD. Feasibility and acceptability of C-PRIME: A health promotion intervention for family caregivers of patients with colorectal cancer. Support Care Cancer. 2024 Feb 28;32(3):198. doi: 10.1007/s00520-024-08395-5. PMID 38416143